CLINICAL TRIAL: NCT01943721
Title: A Study of the VISION5 Product in Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ForSight Vision5, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ForSight VISION5 Study 504
Record Dates: First submitted 2013-09-10; First posted 2013-09-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Ocular Hypertension; Primary Open Angle Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VISION5 Product (Experimental): VISION5 Product in both eyes
  Interventions: Drug: VISION5 Product

INTERVENTIONS:
Drug: VISION5 Product

SUMMARY:
The objective of this Phase 1 study is to evaluate the VISION5 Product's safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Primary open-angle glaucoma or ocular hypertension in both eyes
* Best-corrected distance vision of 20/100 or better
* Stable visual field

Exclusion Criteria:

* Cup-to-disc ratio greater than 0.8
* Laser surgery for glaucoma/ocular hypertension on one or both eyes within the last 12 months
* Corneal refractive surgery within prior 6 months
* Past history of any incisional surgery for glaucoma at any time
* Corneal abnormalities that would interfere with tonometry readings
* Current participation in an investigational drug or device study or participation in such a study within 30 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Ocular Tonometry (change from baseline) | Week 2, 6, 12 and Months 4,5,6

SECONDARY OUTCOMES:
Safety as assessed by Slit Lamp Exam | Weeks 2,6,12 and Months 4,5,6

CONTACTS AND LOCATIONS:
Overall Officials: Anne Rubin, Study Director — ForSight VISION5
Locations (1):
- Contact ForSight VISION5 for Trial Locations, Contact ForSight Vision5 For Trial Locations, Latvia